CLINICAL TRIAL: NCT00363233
Title: The Effects of Flax Lignans on Lipid Profile and Glucose Management in Type 2 Diabetes: a Randomized Double-Blind Cross-Over Study
Brief Title: The Potential Effects and Mechanisms of Flax Lignans on Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 04DZ14007
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2007-01-09 (Estimated); Status verified 2007-01

CONDITIONS: Type 2 Diabetes; Hypercholesterolemia
Keywords: type 2 diabetes; lignans; flaxseed; cholesterol
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypercholesterolemia

INTERVENTIONS:
Drug: flax lignans

SUMMARY:
The purpose of the study is to improving the lipid profile and glucose control in type 2 diabetic patients with supplementation of flax lignans. We hypothesize that flax lignans supplement will improve the cholesterol profile and glucose control in type 2 diabetic patients.

DETAILED DESCRIPTION:
The prevalence of type 2 diabetes is increasing dramatically in the last decade in China. Hyperlipidemia is a comorbid condition in type 2 diabetes and increase the adverse health outcomes. Flax lignans, a phytoestrogen found in flaxseed is thought to be the compound responsible for cholesterol-lowering effect of flaxseed. Our purpose is to improving the lipid profile in type 2 diabetic patients with supplementation of flax lignans.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed type 2 diabetes
* Age: 50-79 years old
* LDL-cholesterol more than 2.9 mmol/l

Exclusion Criteria:

* Current or previous (within 6 months) use of estrogen therapy
* Cancer
* Chronic gastrointestinal diseases
* Current use of antibiotics
* Any severe liver or renal diseases
* Systolic blood pressure more than 180 mmHg or phase 3 hypertension
* Any severe mental diseases
* Severe cardio- or cerebro-vascular diseases

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2006-03; Study Completion 2006-12

PRIMARY OUTCOMES:
Total cholesterol at 3 months

SECONDARY OUTCOMES:
LDL and triglycerides at 3 months; Blood glucose and HbA1C at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Xu Lin, MD, PhD, Principal Investigator — Institute for Nutritional Sciences, Chinese Academy of Sciences
Locations (1):
- Institute for Nutritional Sciences, Chinese Academy of Sciences; Huadong Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Pan A, Sun J, Chen Y, Ye X, Li H, Yu Z, Wang Y, Gu W, Zhang X, Chen X, Demark-Wahnefried W, Liu Y, Lin X. Effects of a flaxseed-derived lignan supplement in type 2 diabetic patients: a randomized, double-blind, cross-over trial. PLoS One. 2007 Nov 7;2(11):e1148. doi: 10.1371/journal.pone.0001148. PMID 17987126